CLINICAL TRIAL: NCT05347628
Title: A Phase I, Open-label, Multicenter, Dose Escalation and Dose Expansion Study to Assess the Safety, Tolerability, Pharmacokinetics and Anti-tumor Efficacy of PLB1004 in Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Assessing the Safety and Efficacy of PLB1004 in Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Avistone Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLB1004-I-01
Record Dates: First submitted 2022-04-13; First posted 2022-04-26 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-07

CONDITIONS: Non-Small-Cell Lung Cancer
Keywords: Non-Small-Cell Lung Cancer; EGFR; NSCLC; Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PLB1004 (Experimental): PLB1004 given alone as monotherapy.
  Interventions: Drug: PLB1004

INTERVENTIONS:
Drug: PLB1004 — PLB1004 is a capsule in the form of 10mg and 40mg.

SUMMARY:
This is a phase I, open-label, multicenter study to assess the safety, tolerability, pharmacokinetics and preliminary antitumor activity of PLB1004, and to determine the maximum tolerated dose (MTD), dose-limiting toxicities (DLTs) and recommended phase II dose (RP2D).

DETAILED DESCRIPTION:
The study includes a Dose-escalation Part and a Dose Expansion Part. The aim of the Dose-escalation Part is to estimate the MTD (if possible), identify the DLT (if possible) and the RP2D for PLB1004. The Dose Expansion Part is to further assess the clinical efficacy and safety of PLB1004.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and the willingness to sign a written informed consent document；
2. Aged at least 18 years old;
3. Histologically or cytologically confirmed advanced non-small cell lung cancer;
4. Patients with EGFR or HER2 mutations;
5. ECOG Performance Status of 0-2;
6. Life expectancy is not less than 12 weeks;
7. At least one measurable lesion as defined by RECIST1.1;

Exclusion Criteria:

1. For the Dose Expansion Part: Patients who have received prior treatment with Poziotinib or TAK788 or other EGFR/HER2 exon20 insertion inhibitors should be excluded；
2. Any cytotoxic drugs or other anticancer drugs from a previous treatment regimen within 14 days prior to the first dose of PLB1004；
3. Major surgery (e.g., intra-thoracic, intra-abdominal or intra-pelvic) within 4 weeks prior (2 weeks for resection of brain metastases) to starting PLB1004 or who have not recovered from side effects of such procedure;
4. Thoracic radiotherapy to lung fields ≤ 4 weeks prior to starting PLB1004. For all other anatomic sites (including radiotherapy to thoracic vertebrae and ribs), radiotherapy ≤ 2 weeks prior to starting PLB1004 or patients who have not recovered from radiotherapy-related toxicities. Palliative radiotherapy for bone lesions ≤ 2 weeks prior to starting PLB1004 is allowed;
5. Patients receiving treatment with medications that meet one of the following criteria and that cannot be discontinued at least 1 week prior to the start of treatment with PLB1004 and for the duration of the study:

   * Strong inhibitors of CYP3A4
   * Strong inducers of CYP3A4
   * Inducers or inhibitors of P-gp
6. Patients with symptomatic central nervous system (CNS) metastases who are neurologically unstable or have required increasing doses of steroids within the 2 weeks prior to study entry to manage CNS symptoms;
7. Clinically significant, uncontrolled heart diseases;
8. Presence or history of a malignant disease other than NSCLC that has been diagnosed and/or required therapy within the past 3 years. Exceptions to this exclusion include the following: completely resected basal cell and squamous cell skin cancers, indolent malignancies that currently do not require treatment, and completely resectedcarcinoma in situ of any type;
9. Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease;
10. History of hypersensitivity to active or inactive excipients of PLB1004 or drugs with a similar chemical structure or class to PLB1004;
11. Pregnant or nursing women;
12. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Estimated)
Dates: Start 2020-08-25 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs) | 2 years
  A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
DLTs of Orally Administered PLB1004 | 28 days
  Toxicity will be evaluated according to the NCI CTCAE, Version 5.00. DLT will be defined as any of the events specified in the protocol that are considered by the investigator to be at least possibly related to therapy with study medications.
Maximum Tolerated Dose (MTD) of Orally Administered PLB1004 | 28 days
  The MTD is the highest dose level at which the participant tolerates treatment without dose-limiting toxicities.
Recommended Phase II Dose (RP2D) of Orally Administered PLB1004 | 2 years
  The RP2D is the maximum tolerated dose (MTD) or less. An RP2D less than the MTD may be chosen if aspects of tolerability or efficacy not encompassed by the MTD determination suggest utilizing a lower dose.

SECONDARY OUTCOMES:
Area Under the Curve (AUC) of PLB1004 | Up to approximately 28 days; Pre-dose and multiple time points post-dose
  The AUC values are based on the plasma concentration-time profile of PLB1004. To characterize the pharmacokinetics of PLB1004.
Maximum plasma concentration (Cmax) of PLB1004 | Up to approximately 28 days; Pre-dose and multiple time points post-dose
  The Cmax values are based on the plasma concentration-time profile of PLB1004. To characterize the pharmacokinetics of PLB1004.
Time to maximum plasma concentration (Tmax) of PLB1004 | Up to approximately 28 days; Pre-dose and multiple time points post-dose
  The Tmax values are based on the plasma concentration-time profile of PLB1004. To characterize the pharmacokinetics of PLB1004.
Overall Response Rate (ORR) | 3 years
  ORR is defined as the proportion of subjects with confirmed best overall response of complete response (CR) or partial response (PR) according to RECIST 1.1.
Progression-Free Survival (PFS) | 3 years
  PFS is defined as the time interval from the date of starting treatment until the first date at which the criteria for progressive disease (PD) according to RECIST 1.1 are met or death, whichever occurs first.
Overall Survival (OS) | 3 years
  OS is defined as the time from date of starting treatment to date of death due to any cause.
Disease Control Rate (DCR) | 3 years
  DCR is defined as the percentage of participants who have achieved CR, PR, or SD after the initiation of study drug.
Duration of Response (DOR) | 3 years
  DOR is defined as the time from first documented response of CR or PR to date of first documented progression or death according to RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wu, MD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No